CLINICAL TRIAL: NCT02577588
Title: Phase I Trial of Adoptive T Cell Therapy With Activated P53 Specific T Cells for Treatment of Advanced Colorectal Cancer
Brief Title: Trial of Adoptive T Cell Therapy With Activated P53 Specific T Cells for Treatment of Advanced Colorectal Cancer
Acronym: ATACC
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: not feasible
Sponsor: National Center for Tumor Diseases, Heidelberg (Other)
Collaborators: German Cancer Research Center (Other); University Hospital Heidelberg (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCT-2009-11-03-1055
Record Dates: First submitted 2015-05-06; First posted 2015-10-16 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2018-03

CONDITIONS: Colorectal Carcinoma
Keywords: p53 Antigen; T cell therapy; autologous; Adoptive Cellular Immunotherapy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- re-activated T cells (Experimental): Ten patients with CRC stage UICC IV under routine first line FOLFOX 6/Bevacizumab therapy are planned to receive a singular treatment with an autologous T cell product at a dose of 5x10^7 (first three or six patients) or 5x10^8 (last four or seven patients) cells.
  Interventions: Biological: re-activated T cells

INTERVENTIONS:
Biological: re-activated T cells — autologous reactivated T cells against p53
  Other Names: autologous T cells; p53 activated T cells

SUMMARY:
The study "Phase I trial of Adoptive T cell Therapy with Activated P53 specific T cells for Treatment of Advanced Colorectal Cancer" is an open label, single arm trial.

DETAILED DESCRIPTION:
Most patients with colorectal carcinoma (CRC) accumulate high numbers of endogenous tumor antigen specific cytotoxic and helper memory T cells in their blood. Upon appropriate reactivation, tumor antigen specific T cells can recognize and eliminate autologous tumor cells. This can be achieved ex vivo by their stimulation with antigen pulsed autologous dendritic cells in the absence of regulatory T cells. Upon adoptive transfer, specifically reactivated T cells from cancer patients can efficiently reject autologous human tumors in vivo.

A major target antigen of anti tumor effector T cells in CRC patients is p53, which is overexpressed in many colorectal cancers. Within this clinical trial, high numbers of endogenous tumor specific T cells will be harvested by leukapheresis from the blood of CRC patients harbouring p53-reactive T cells. Isolated T cells will be depleted from regulatory T cells and specifically reactivated for three days ex vivo with three synthetic long peptides containing the most immunogenic regions of p53 using autologous dendritic cells as antigen presenting cells. Activated T cells will be re-infused into the patients.

Ten patients with CRC stage UICC IV under routine first line FOLFOX 6/Bevacizumab therapy are planned to receive a singular treatment with an autologous T cell product at a dose of 5x10^7 (first three or six patients) or 5x10^8 (last four or seven patients) cells.

Patient treatment and follow-up will be performed at the National Center for Tumor Diseases (NCT) and at the Department of General, Visceral and Transplantation Surgery, University of Heidelberg. Leukapheresis will take place at the DRK-Blutspendedienst Baden-Württemberg-Hessen in Mannheim and generation of therapeutic cells will be performed at the GMP Unit Cellular Therapy of the DKFZ. Analysis of blood samples with respect to special immune parameters is carried out at the Immune Monitoring Laboratory, Department of Translational Immunology at the NCT, Heidelberg.

The primary objective of this study is to evaluate the safety and tolerability of an adoptive transfer of ex vivo reactivated p53 specific T cells obtained from peripheral blood.

ELIGIBILITY:
Inclusion Criteria

* Histologically confirmed UICC stage IV colorectal cancer and non resectable primary tumor and/or metastases
* Previous palliative standard systemic treatment with FOLFOX, FOLFIRI, or FOLFIRINOX in combination with Bevacizumab or Cetuximab/Panitumumab, and currently under respective treatment
* The following situation after at least four cycles with FOLFOX, FOLFIRI, or FOLFIRINOX in combination with Bevacizumab or Cetuximab/Panitumumab should apply:

  * Disease control (stable disease, partial response or complete response) according routine imaging
  * Resection of tumor and/or metastases still impossible
  * Tolerability of systemic treatment
  * The decision of the treating physician is to continue the standard background treatment
* Presence of tumor-reactive T cells in the blood as detected by ex vivo IFN-γ EliSpot assay and classification of the reaction as a response in a blood sample
* ECOG-performance status 0 or 1
* Adequate vein status at both cubital fossas for 16 G puncture (white permanent venous catheter, Braunüle; EN ISO 6009)
* Age ≥ 18 years, any ethnic origin and gender
* Ability of the patient to understand the character and individual consequences of the clinical trial
* Patients should be willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures
* Written informed consent (must be available before enrolment in the trial)
* Negative pregnancy test (females of childbearing potential)
* Women with childbearing potential and male patients with partners of childbearing potential should be willing to use adequate contraception (failure rate less than 1% per year when used consistently and correctly) during the study and three month last application of T cell therapy
* At the screening visit the following laboratory parameters apply and should be within the ranges specified:

Lab Parameter Range WBC ≥4000/mm3 (≥4000/ul) Platelets ≥80.000/mm3 (≥80.000/ul) Creatinine ≤1.5mg/dl ALT, AST, and total bilirubin < 2.5 x ULN HB* > 9 g/dl

*HB is controlled again at day -11 at DRK Mannheim as part of the procedures before leukapheris.

Exclusion Criteria

* Brain or leptomeningeal metastases, shown by MRI Scan during Screening phase or by routinely available other appropriate diagnostic (CT, MRI, PET) conducted within 3 months prior to inclusion.
* Previous malignancy within the past 5 years. However: Patients who had curatively treated basal cell carcinoma of the skin, early gastrointestinal cancer treated by endoscopic resection and/or in situ carcinoma of the cervix are allowed for enrolment.
* History of organ allograft or prior hematopoetic stem cell transplantation
* History of inflammatory bowel disease (ulcerative colitis, Crohn's disease)
* History of symptomatic autoimmune disease (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [e.g., Wegener's Granulomatosis])
* History of motor neuropathy considered of autoimmune origin (e.g., Guillain-Barré Syndrome)
* Clinically significant cardiac disease (NYHA Class III or IV).
* Other serious illnesses, which renders the patient unsuitable for study entry or multiple blood sampling
* Serious intercurrent illness, requiring hospitalization
* HIV and/or HBC/HCV positivity, tested by appropriate infection diagnostics during screening period
* Any active infection or signs or symptoms of infection
* Patient pregnant or breastfeeding
* History of hypersensitivity to the investigational medicinal product or to any excipient present in the investigational medicinal product or to anti-coagulance auxiliary medicianal product (Heparin prophylaxis)
* Treatment with immunosuppressive drugs (e.g. systemic corticosteroids) besides intermittent, anti-emetic steroid application during treatment with FOLFOX, FOLFIRI, or FOLFIRINOX in combination with Bevacizumab or Cetuximab/Panitumumab. Topical or inhalation steroids are permitted.
* Treatment with any approved anti-cancer therapy within 28 days prior to enrolment, except the background treatment FOLFOX, FOLFIRI, or FOLFIRINOX in combination with Bevacizumab or Cetuximab/Panitumumab.as recommended by that trial protocol
* Treatment with any live attenuated vaccine within 4 weeks before first administration of investigational medicinal product
* Treatment with any other investigational agent or participation in another interventional clinical trial within 28 days prior to enrolment.

No patient will be allowed to enroll in this trial more than once.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2018-02-19 (Actual); Study Completion 2018-02-19 (Actual)

PRIMARY OUTCOMES:
Safety | 45 days
  The primary endpoint is the Dose Limiting Toxicity (DLT), defined as: any adverse event (AE) ≥ Grade 3 according to the Common Terminology Criteria for Adverse Events (CTCAE version 4.03), that is judged by the investigator as definitely, probably or possibly related to the investigational medicinal product (IMP) or to the combination of the IMP and the treatment with FOLFOX 6/Bevacizumab.

SECONDARY OUTCOMES:
evaluation of p53 specific T cell Responses by analysing data from EliSpot assay | day 0, 10, 17, 24, 31
  The response of a patient to the p53 peptide mix or to each of the single p53 peptides

CONTACTS AND LOCATIONS:
Overall Officials: Alexis Ulrich, MD Prof. Dr., Principal Investigator — University Hospital Heidelberg
Locations (1):
- National Center for Tumor desease NCT, Heidelberg, Baden-Wurttemberg, Germany